CLINICAL TRIAL: NCT00006274
Title: Study of Energy Requirements in Critically Ill Newborns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Indiana University School of Medicine (Other)
Other Study IDs: NCRR-M01RR00750-9044; IU-9703-22
Record Dates: First submitted 2000-09-11; First posted 2000-09-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Respiratory Distress Syndrome
Keywords: cardiovascular and respiratory diseases; neonatal disorders; rare disease; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Tract Diseases; Infant, Newborn, Diseases; Rare Diseases

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
OBJECTIVES:

I. Determine the total energy expenditure in term and preterm infants in both well and ill states using the doubly labeled water method.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are assigned to one of three groups according to gestational age (24-28 weeks estimated gestational age (EGA) vs 29-34 weeks EGA vs 35 weeks EGA and over) and severity of respiratory illness (need for high frequency ventilation vs stable conventional ventilator settings or extubated within past 24 hours vs no need for mechanical ventilation).

Patients receive water labeled with deuterium and oxygen O 18 by mouth or by gastrostomy tube on days 1 and 7. Urine samples are collected prior to the first dose, 4-6 hours after the first dose, and then every 24 hours until the second dose. All urine is collected for 4-6 hours after the second dose. Samples are analyzed by dual inlet isotope ratio mass spectrometry.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Infants with estimated gestational age (EGA) of at least 24 weeks with respiratory illness who are on high frequency ventilation (HFOV) and meet the following conditions: Appropriate size for gestational age (AGA) No congenital anomalies No medical complications, including seizures and necrotizing enterocolitis

OR

Control infants with EGA of at least 24 weeks Must meet 1 of the following conditions: Requirement for stable conventional ventilator settings with respiratory index score of less than 2.5 and/or extubated within past 24 hours No requirement for mechanical ventilation Must meet all of the following conditions: AGA No congenital anomalies No medical complications, including seizures and necrotizing enterocolitis No documented sepsis by positive blood culture No supplemental oxygen use (infants 35 weeks EGA and over only)

--Prior/Concurrent Therapy--

HFOV group: Concurrent surfactant, theophylline, or inotrope (vasopressor) therapy allowed

Control group: No concurrent inotrope (vasopressor) therapy

Ages: 24 Hours to 120 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 1997-03

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A. Leitch, Study Chair — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States